CLINICAL TRIAL: NCT06119334
Title: Promoting Healthy Exercise to Conscientious Christians
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: York University (Other)
Responsible Party: Principal Investigator, Paul Ritvo, Principal Investigator, York University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3835
Record Dates: First submitted 2023-07-09; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Sedentary Behavior
Keywords: internet-based intervention with health coaching;
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Paralell group design with intervention participants compared to wait-list control subjects. 16 weeks intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Sixteen weeks of phone-based counselling at a rate of 1 session/week and ongoing access to a online platform (Nex J Connected Wellness) that has health promotion text and videos readily accessed in combination with text messaging exchanges between counselor and participant. Participants receive a Fitbit which is connected to the Nex J Connected Wellness such that counselors can monitor steps/day.
  Interventions: Behavioral: Online intervention
- Wait list control (No Intervention): Participants wait for 16 weeks.

INTERVENTIONS:
Behavioral: Online intervention — Phone counselling for 1 hour/week over 16 weeks and access to the online platform with health promotion materials (videos, text, audios)
  Arms: Experimental

SUMMARY:
Given the importance of reducing mortality-morbidity, more effective Physical Activity (PA) interventions are important, and the recently observed stabilizations of PI levels suggest that novel methods must be explored (Ozemek et al., 2019).

This study aims to provide a select sedentary subpopulation with a customized intervention hypothesized to increase their PA adoption. Novel recruiting methods are used to identify a target subpopulation (based on multiple characteristics) that can be contacted in multiple sections of North America. We will intervene online and rigorously test the theoretical formulations that identify the subpopulation and the customized intervention.

DETAILED DESCRIPTION:
Physical inactivity (PI) in North America (NA) is associated with high levels of excess morbidity-mortality (Arraiz et al., 1992; Knight, 2012; Villeneuve et al., 1998) with significant decreases in morbidity-mortality predicted with increased physical activity (PA) in recent literature (del Pozo Cruz, et al., 2022; Fogelholm, 2010; Katzmarzyk & Mason, 2009; Peterson et al., 2014; Warburton & Bredin, 2017). The lower range of prevalence indicators of PI suggest that 47% of Americans (Centers for Disease Control and Prevention [CDC], n.d.) and 51% of Canadians (Statistics Canada, 2021) do not reach the PA guidelines of 150 minutes of moderate-to-vigorous physical activity (MVPA) weekly. The upper end estimates point to approximately 80% of adults being too sedentary to gain health benefits (Piercy et al., 2018). Recent evidence analyzed by the US 2018 Physical Activity Guidelines Advisory Committee (US Department of Health and Human Services [HHS], 2018), based on extensive literature review, indicates strong PI associations with increased all-cause mortality. Also noteworthy were specifically increased incidences of: 9.9% for cardiovascular diseases; 6.5% for stroke; 2.2% for hypertension; and 5.9% for Type 2 diabetes. Increased incidences were also associated with cancer-related diseases (2.9% for bladder cancer; 3.6% for breast cancer; and 3.9% for colon cancer) (Katzmarzyk et al., 2022). The estimated healthcare costs attributable to PI in Canada were $2.1 billion (1999) and $2.4 billion (2009), the latter figure associated with indirect costs of $4.3 billion and total costs of $6.8 billion (Katzmarzyk et al., 2000). Given the importance of reducing mortality-morbidity, more effective Physical Activity (PA) interventions are important, and the recently observed stabilizations of PI levels suggest that novel methods must be explored (Ozemek et al., 2019). This study aims to provide a select sedentary subpopulation with a customized intervention hypothesized to increase their PA adoption. Novel recruiting methods are used to identify a target subpopulation (based on multiple characteristics) that can be contacted in multiple sections of North America. We will intervene online and rigorously test the theoretical formulations that identify the subpopulation and the customized intervention.

Physical inactivity (PI) in North America (NA) is associated with high levels of excess morbidity-mortality (Arraiz et al., 1992; Knight, 2012; Villeneuve et al., 1998) with significant decreases in morbidity-mortality predicted with increased physical activity (PA) in recent literature (del Pozo Cruz, et al., 2022; Fogelholm, 2010; Katzmarzyk & Mason, 2009; Peterson et al., 2014; Warburton & Bredin, 2017).

The lower range of prevalence indicators of PI suggest that 47% of Americans (Centers for Disease Control and Prevention [CDC], n.d.) and 51% of Canadians (Statistics Canada, 2021) do not reach the PA guidelines of 150 minutes of moderate-to-vigorous physical activity (MVPA) weekly. The upper end estimates point to approximately 80% of adults being too sedentary to gain health benefits (Piercy et al., 2018).

Recent evidence analyzed by the US 2018 Physical Activity Guidelines Advisory Committee (US Department of Health and Human Services [HHS], 2018), based on extensive literature review, indicates strong PI associations with increased all-cause mortality. Also noteworthy were specifically increased incidences of: 9.9% for cardiovascular diseases; 6.5% for stroke; 2.2% for hypertension; and 5.9% for Type 2 diabetes. Increased incidences were also associated with cancer-related diseases (2.9% for bladder cancer; 3.6% for breast cancer; and 3.9% for colon cancer) (Katzmarzyk et al., 2022). The estimated healthcare costs attributable to PI in Canada were $2.1 billion (1999) and $2.4 billion (2009), the latter figure associated with indirect costs of $4.3 billion and total costs of $6.8 billion (Katzmarzyk et al., 2000).

Given the importance of reducing mortality-morbidity, more effective Physical Activity (PA) interventions are important, and the recently observed stabilizations of PI levels suggest that novel methods must be explored (Ozemek et al., 2019). This study aims to provide a select sedentary subpopulation with a customized intervention hypothesized to increase their PA adoption. Novel recruiting methods are used to identify a target subpopulation (based on multiple characteristics) that can be contacted in multiple sections of North America. We will intervene online and rigorously test the theoretical formulations that identify the subpopulation and the customized intervention.

Aims and Objectives:

A. To estimate the approximate number of North American individuals who visit Christian - oriented online programs and dialogue on these programs about personally meaningful issues. This estimate is relevant to the potential for online PA interventions to reach ample populations and deliver adoption stimulating, reinforcing effects that result in increased MVPA.

B. To assess within a randomized controlled trial (RCT) whether an online Christianbased CBT-PA intervention is more effective than a comparison wait list control condition, in terms of increased MVPA as assessed by self-report (IPAQ), Fitbit (online] tracked steps, and self-reported changes in body mass index (BMI).

C. To assess within a RCT whether engagement with and/or adherence to the online Christian-based PA intervention (i.e. online workbooks completed, online text messages exchanged, phone sessions completed) predicts increased MVPA.

D. To compare the cost-effectiveness of the online Christian-based PA intervention to the comparison wait-list control condition at post-intervention (4 months) and at 2 months post-follow up (6 months).

Hypotheses

A. An increasing number of North Americans visit Christian online groups and programs and exchange dialogues on personally meaningful Christianity issues. Amidst the ~231 million Christians estimated to reside in North America, we believe an increasing proportion (30% to 40%) are engaging in online visits per month (Johnson et al., 2018).

B. The Christian-based CBT-PA intervention is more effective than the comparison (wait list control) condition in terms of significantly increased MVPA as assessed by self-report (IPAQ), Fitbit (online) tracked steps, and self-reported changes in body mass index (BMI).

C. Engagement in and adherence to the online Christian-based PA intervention (i.e. online workbooks completed, online text messages exchanged, phone sessions completed) will predict significantly increased MVPA in the experimental group.

D. The online Christian-based PA intervention program will be significantly more cost effective when compared to the comparison condition at postintervention and at 2 months follow up.

ELIGIBILITY:
Inclusion Criteria:

(1) 25 to 55 years old; (2) self-identification as a regular church attendee (Lazerwitz, 1962); (3) willingness to complete the Big Five Inventory (BFI) (John et al., 2008; John & Srivastava, 1999; (4) BFI scores that are 1 SD > the mean score typically derived in most published studies; (5) willingness to receive and use a loaned Fitbit Versa 2 delivered by FedEx and commit to wearing it during daytime hours on a daily basis for the duration of the 16 week intervention (6) BMI between 27 and 33; (7) fluent in English; (8) approval from a primary care physician for initiating a graded-incremental walking exercise routine; (9) ability to walk for 30 minutes at a time without significant self-identification of pain and/or orthopedic dysfunction.

Exclusion Criteria: 1) Individuals who self-report a past or present diagnosis of Bipolar Disorder, Borderline Personality Disorder, Obsessive-Compulsive Disorder, Schizophrenia, Substance Abuse/Addiction in the past three months will be excluded; suicidal ideation or attempted suicide in the past six months prior to the study are also exclusion factors; (2) individuals with a self-reported co-morbid illness or condition that could be negatively affected by walking exercise; 3) individuals who report walking 20 minutes per day (on average) or more.

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-11-25 (Estimated); Primary Completion 2025-11-10 (Estimated); Study Completion 2025-12-09 (Estimated)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) (low-moderate-high) | Baseline
  Self report of physical activity reflecting current activity
International Physical Activity Questionnaire (IPAQ) (low-moderate-high) | 8 weeks
  Change in self report of physical activity
International Physical Activity Questionnaire (IPAQ) (low-moderate-high) | 16 weeks
  Change in self report of physical activity
Fitbit Versa 2 Fitness Tracker connected to the NexJ Connected Wellness platform. | 8 weeks
  Electronic monitoring of steps
Fitbit Versa 2 Fitness Tracker connected to the NexJ Connected Wellness platform. | 16 weeks
  Change in Electronic monitoring of steps

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Baseline
  Weight and height measurements
Body Mass Index (BMI) | 16 weeks
  Change in Weight and height measurements
Patient Health Questionnaire-9 (PHQ - 9) (0-27) | Baseline
  Brief Measure of Depression
Patient Health Questionnaire-9 (PHQ - 9) (0-27) | 16 weeks
  Change in Brief Measure of Depression
General Anxiety Disorder-7 (GAD-7) (0-21) | Baseline
  Brief measure of Anxiety
General Anxiety Disorder-7 (GAD-7) (0-21) | 8 weeks
  Change in Brief measure of Anxiety
General Anxiety Disorder-7 (GAD-7) (0-21) | 16 weeks
  Change in Brief measure of Anxiety
Duke University Religion Index (DUREL) (5-27) | Baseline
  Religious committment
Duke University Religion Index (DUREL) (5-27) Duke University Religion Index | 8 weeks
  Change in Duke University Religion Index
Duke University Religion Index (DUREL) (5-27) Duke University Religion Index (5-27) | 16 weeks
  Change in Duke University Religon Index
Quality of life (EQ-5D) (0-100) | Baseline
  Utility-based measure
Quality of life (EQ-5D) (0-100) | 8 weeks
  Change in Quality of life (EQ-5D)
Quality of life (EQ-5D) (0-100) | 16 weeks
  Change in Quality of life (EQ-5D)
12 item Grit Scale (12-60) | Baseline
  Measure of 'grit' - long term passionate committment
12 item Grit Scale (12-60) | 8 weeks
  Change in 12 item Grit Scale
12 item Grit Scale (12-60) | 16 weeks
  Change in 12 item Grit Scale
  Change in
  Change in Measure of 'grit' - long term passionate committment

CONTACTS AND LOCATIONS:
Locations (1):
- York University - School of Kinesiology and Health Science, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Posting on website
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2023-2025 - 2 years
Access Criteria: all interested investigators